CLINICAL TRIAL: NCT03765047
Title: A Rigorous Evaluation of the Relationship Between Physical Activity and Education Outcomes in Georgia's Elementary Schools (RWJF)
Brief Title: A Rigorous Evaluation of the Relationship Between Physical Activity and Education Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Julie A Gazmararian, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00095600; 74281 (Other Grant/Funding Number: Robert Wood Johnson Foundation)
Record Dates: First submitted 2018-12-03; First posted 2018-12-05 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Physical Activity
Keywords: Standardized Test Score; Academic Achievement
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): This study arm includes the schools where the School Team (school teachers, coordinator) receives the physical activity intervention. The intervention consists of four parts:
  1. School Engagement and Assessment
  2. Training
  3. Physical Activity Equipment and Resources
  4. Ongoing Assessment and Technical Assistance
  Interventions: Behavioral: Intervention Arm
- Control Arm (No Intervention): The control arm includes the schools where the School Team does not receive any intervention but all the necessary data will be collected.

INTERVENTIONS:
Behavioral: Intervention Arm — The physical activity intervention consists of:
  1. School Engagement and Assessment - Based on the customized assessment, training is provided for school staff to develop the capacity to increase PA. A school PA team is established.
  2. Training - School teams are provided with ongoing in-person and virtual training to learn strategies for increasing PA before and during the school day. A training summit meeting will occur each summer, starting with the summer prior to the intervention. Teams will create a weekly calendar of activities to increase PA time to a minimum of 40 mts/day.
  3. PA Equipment and Resources - After training, schools are provided with PA equipment, resources and teaching aids to facilitate the integration of PA into the school day.
  4. Ongoing Assessment and Technical Assistance - Student accelerometer data will allow for monitoring of PA levels, so that additional technical assistance for classroom teachers can be provided if needed
  Arms: Intervention Arm

SUMMARY:
The study is a prospective study to examine the impact of a school-based physical activity intervention on fourth and fifth grade elementary students' academic achievement, as measured by standardized test scores.

DETAILED DESCRIPTION:
Serving more than 95% of US children ages 5-17, the school environment is a valuable setting to engage students in Physical Activity (PA) through the day, but is limited when physical education programs have insufficient curricular, time, financial and staffing allocations. A growing body of research supports the premise that interventions focused on increasing physical activity in schools may be more successful if supported by evidence that increased PA improves academic achievement, that is the clear priority for limited school time and resources.

The purpose of this study is to examine the impact of a school-based physical activity intervention on fourth and fifth grade elementary students' academic achievement, as measured by standardized test scores. Baseline information about current physical activity practices will be collected. Schools will receive ongoing in-person and virtual training, and schools will be provided physical activity equipment, resources, and teaching aids. Student accelerometer data will allow for monitoring of physical activity levels. This study seeks to address gaps in the literature by studying the efficacy of a well-established intervention that has been shown to impact school physical activities practices, and shows promise of efficacy for improving student education outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 4th grade students from the elementary schools in the Gwinnett County district

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4968 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2020-06-19 (Actual); Study Completion 2020-06-19 (Actual)

PRIMARY OUTCOMES:
Change in the Georgia Milestones standardized test scores in math | Up to 2 years
  The Georgia Milestones comprehensive summative assessment is administered annually in the spring for students in grades 3 to 8. The test was first used in Spring 2015 and is the best objective universal indicator of students' academic performance in Georgia. Georgia Milestones measures how well students have learned the knowledge and skills outlined in the state-adopted content standards in English language arts, mathematics, science, and social studies. The tests are scored with four achievement levels. Level 1: Beginning Learner, Level 2: Developing Learner, Level 3: Proficient Learner, and Level 4: Distinguished Learner. For grade 3 the scores for the different levels of math are 290-474, 475-524, 525-579, and 580-705; for grade 4, 270-474, 475-524, 525-584, and 580-715; for grade 5, 265-474, 475-524, 525-579, and 580-725, respectively. The scores from the 3rd grade (pre-intervention) are compared to scores at the end of 4th and 5th grades.
Change in the Georgia Milestones standardized test scores in reading | Up to 2 years
  The Georgia Milestones comprehensive summative assessment is administered annually in the spring for students in grades 3 to 8. The test was first used in Spring 2015 and is the best objective universal indicator of students' academic performance in Georgia. Georgia Milestones measures how well students have learned the knowledge and skills outlined in the state-adopted content standards in English language arts, mathematics, science, and social studies.The tests are scored with 4 achievement levels. Level 1: Beginning Learner, Level 2: Developing Learner, Level 3: Proficient Learner, and Level 4: Distinguished Learner. For grade 3 the scores for the different levels for reading are 180-474, 475-524, 525-580, and 581-830; for grade 4, 210-474, 475-524, 525-573, and 574-775; for grade 5, 210-474, 475-524, 525-586, and 587-760, respectively. The scores from the 3rd grade assessment (pre-intervention) are compared to scores at the end of 4th and 5th grades.

SECONDARY OUTCOMES:
Change in the Lexile/reading level for language arts | Up to 2 years
  Lexile Level is a popular method used by schools to measure a student reader's ability. It serves two unique functions: it is a measure of how difficult a text is, and a measurement of a student's reading ability level. A student receives his or her Lexile measure by taking a school-administered Scholastic Reading Inventory test, which is specifically designed to measure Lexile or reading ability, or by taking a standardized reading test which converts the reader's results to a Lexile measure. The normal Scholastic Guided Reading Lexile ranges for 3rd grade are 100-1120, 180-1280 for 4th grade, and 330-1280 for 5th grade.
Change in the class grades for reading | Up to 2 years
  Class grades are calculated from the reading tests administered during the school year. The class grades for reading from 3rd grade are compared to 4th and 5th grades, and class reading grades are also compared between the students in the intervention arm and control arm.
Change in the class grades for math | Up to 2 years
  Class grades are calculated from the math tests administered during the school year. The class math grades from 3rd grade are compared to 4th and 5th grades, and math grades are also compared between the students in the intervention arm and control arm.
Number of Disciplinary Referrals | Up to 2 years
  Disciplinary referrals collected by teachers (including information regarding incident date, incident type, action taken, rule number broken, and discipline code) will be compared between grade levels and also compared between the students in the intervention arm and control arm.
Number of days of absence | Up to 2 years
  The number of days that students were absent from school during the academic year will be collected from school records and compared between grade levels and also compared between the students in the intervention arm and control arm.
Number of days a student was tardy to the school | Up to 2 years
  The number of days that students were tardy to school during the academic year will be collected from school records and compared between grade levels and also compared between the students in the intervention arm and control arm.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Gazmararian, PhD/MPH, Principal Investigator — Emory University
Locations (1):
- Gwinnett County Elementary Schools, Lawrenceville, Georgia, United States

REFERENCES:
- [Derived] Behringer HK, Saksvig ER, Boedeker PJ, Elish PN, Kay CM, Calvert HG, Meyer AM, Gazmararian JA. Physical activity and academic achievement: an analysis of potential student- and school-level moderators. Int J Behav Nutr Phys Act. 2022 Aug 30;19(1):110. doi: 10.1186/s12966-022-01348-3. PMID 36042515
- [Derived] Elish PN, Bryan CS, Boedeker PJ, Calvert HG, Kay CM, Meyer AM, Gazmararian JA. The longitudinal association between objectively-measured school-day physical activity and academic achievement in US elementary school students. Int J Behav Nutr Phys Act. 2022 Jul 23;19(1):90. doi: 10.1186/s12966-022-01328-7. PMID 35870926